CLINICAL TRIAL: NCT01733082
Title: The Mycophenolate Pregnancy Registry
Status: Recruiting | Type: Observational
Sponsor: Genentech, Inc. (Industry)
Collaborators: Accord Healthcare, Inc. (Industry); Alkem Laboratories Ltd (Industry); Ascend Laboratories, LLC (Unknown); Amneal Pharmaceuticals, LLC (Industry); Amta labs Limited (Unknown); Apotex Corporation (Unknown); Avet Lifesciences Limited (Unknown); Azurity Pharmaceuticals (Industry); Biocon Pharma Limited (Unknown); Concord Biotech Limited (Unknown); Endo Pharmaceuticals (Industry); Hetero Labs Limited, Unit-V (Unknown); Hikma Pharmaceuticals USA Inc. (Unknown); Hisun Pharmaceuticals (Unknown); Jubilant Cadista Pharmaceuticals, Inc. (Unknown); Lannett Company, Inc. (Industry); Meitheal Pharmaceuticals, Inc. (Unknown); Mylan Pharmaceuticals Inc (Industry); Novartis Pharmaceuticals (Industry); Rising Pharma Holdings, Inc. (Unknown); RK Pharma Inc. (Unknown); Sandoz (Industry); Strides Pharma, Inc (Unknown); Teva Pharmaceuticals USA (Industry); TWi Pharmaceuticals, Inc. (Unknown); VistaPharm, Inc. (Industry); Wuxi Fortune Pharmaceutical Co., Ltd (Unknown); Zydus Pharmaceuticals (Unknown)
Responsible Party: Sponsor
Other Study IDs: ML22679
Record Dates: First submitted 2012-11-20; First posted 2012-11-26 (Estimated); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Heart Transplantation, Kidney Transplantation, Liver Transplantation, Autoimmune Diseases
MeSH Terms: conditions — Autoimmune Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Cohort

SUMMARY:
The Mycophenolate Pregnancy Registry is designed as a prospective, observational registry collecting data regarding mycophenolate exposure during pregnancy, and pregnancy outcomes, fetal and infant outcomes after exposure. Early and later term pregnancy outcomes will be solicited at selected gestational time points. Structural and functional birth defects identified in the perinatal period through one year of life will be collected and classified.

This is a non-proprietary registry and is a component of a comprehensive pregnancy Risk Evaluation and Mitigation Strategy (REMS) plan required by the FDA for all mycophenolate-formulations, including CellCept, Myfortic and any generic formulations.

ELIGIBILITY:
Inclusion Criteria:

* Pregnancy and reported maternal exposure to mycophenolate during pregnancy or within 6 weeks of discontinuing treatment

Exclusion Criteria:

* Pregnancies for which there is paternal exposure only
* Pregnancies occurring outside the U.S.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Pregnancy and reported exposure to mycophenolate during pregnancy or within 6 weeks of discontinuing treatment
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2012-11-20 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Maternal Outcomes: Incidence of Pregnancy Complications | Approximately 13 years
Fetal Outcomes: Incidence of Congenital Disorders | Approximately 13 years
Time/Duration of Mycophenolate Exposure | Approximately 13 years
Mycophenolate Dose/Regimen | Approximately 13 years
Indications for Mycophenolate use | Approximately 13 years
Maternal Medical/Demographic Characteristics | Approximately 13 years

SECONDARY OUTCOMES:
Occurrence of Educational Counseling on the Increased Risks of Birth Defects With Mycophenolate Therapy | Approximately 13 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Genentech, Inc.
Locations (1):
- Quintiles Outcome, Cambridge, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No